CLINICAL TRIAL: NCT05345977
Title: eMotiph: Smart and Innovative E-mental Health Solution to Manage Patients With Schizophrenia
Brief Title: eMotiph: E-mental Health Solution for Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo Pulso (Industry)
Collaborators: Hospital de Sant Pau (Other); Nurogames GmbH (Unknown); Fundació Tic Salut i Social (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 12470-2
Record Dates: First submitted 2022-03-16; First posted 2022-04-26 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia
Keywords: mHealth; Treatment resistent schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: A prospective non-randomised feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unified Protocol (Experimental): The psychotherapy Unified Protocol for Transdiagnostic Treatment of Emotional Disorders.
  Interventions: Device: eMotiph

INTERVENTIONS:
Device: eMotiph — Mobile application for patients with schizophrenia.

SUMMARY:
Although the main objective of current schizophrenia intervention programs is the reduction of symptoms, its rates are around 36%, and recovery rates are 16.5%. Between 30 and 50% of people with schizophrenia obtain little benefit with conventional therapy. They are considered resistant to treatment. Therefore, the development of innovative evidence-based interventions adjunctive to pharmacological and psychological treatment are necessary for improving results in patients with treatment-resistant schizophrenia (TRS). Studies with digital solutions have shown feasibility, acceptability and even preliminary efficacy data. But no earlier published study has focused on TRS.

The eMOTIPH is an innovative solution addressed to TRS and born from the outcomes of the previous study eMOTIPH Part 1 (study of beliefs, needs, and limitations associated with current intervention in TRS patients).

DETAILED DESCRIPTION:
A prospective non-randomised feasibility trial will be performed. People with a diagnosis of treatment-resistant schizophrenia and their informal caregivers will test the digital mental health solution eMOTIPH for 6 months. Psychiatric treatment and psychological intervention (based on the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders; Farchione et al., 2012) will be delivered to patients.

The aim of the study is to evaluate the feasibility, acceptability, usability, satisfaction and perceived quality of life after using the eMOTIPH digital solution.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-55 years old.
* Diagnosis of schizophrenia following the Diagnostic and Statistical Manual of Mental Disorders-5 criteria.
* Meet criteria for treatment-resistant schizophrenia.
* Used to information and communication technology and with the physical capability to use them.

Exclusion Criteria:

* Meet criteria for remission according to the Remission of Schizophrenia Working Group (Andreasen et al., 2005).
* The presence of delusions mainly related to their therapists or with new technologies.
* Hearing, vision or motor impairment that makes it impossible to operate a smartphone.
* Intellectual Developmental Disability.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Technology Acceptance Model Scale (TAM) | Data will be collected immediately after the intervention.
  Degree of acceptance of the digital solution and the intervention delivered. The scale provides scores in 8 dimensions: Perceived Usefulness (score ranges from 5 to 35), Perceived Ease of Use (score ranges from 6 to 42), Attitude (score ranges from 2 to 14), Facilitators (score ranges from 4 to 28), Barriers (score ranges from 2 to 14), Subjective Norm (score ranges from 3 to 21), Intention to Use (score ranges from 1 to 7) and Habits (score ranges from 2 to 14). As much the response trend is located in the positive pole for most of the items, higher acceptability.
User experience questionnaire | Data will be collected immediately after the intervention
  A questionnaire ad hoc will be created where the degree of usability and lived experience after using the digital solution will be measured. This scale has not cut off points. Higher values mean higher usability.
Client Satisfaction Questionnaire (CSQ-8) | Data will be collected immediately after the intervention
  The opinions and conclusions about the digital solution delivered will be asked. The scale has not cut off points. Higher values mean higher satisfaction.

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | Change from Baseline Positive and Negative Syndrome Scale at 6 months.
  Positive, negative and general symptoms of schizophrenia will be assessed. There are not cut off points, direct scores are converted to percentiles. Higher values mean higher presence of positive, negative and general symptoms.
Calgary Depresion Scale for Schizophrenia (CDS) | Change from Baseline Calgary Depresion Scale for Schizophrenia at 6 months.
  The level of depression severity in schizophrenia will be assessed. Cut off points: 0-5, no depression; 6-27, depression.
Beck Anxiety Inventory (BAI) | Change from Baseline Beck Anxiety Inventory at 6 months.
  The level of anxiety will be assessed. The score range is 0-63. A total score of 0-7 is considered minimal range, 8-15 is mild, 16-25 is moderate, and 26-63 is severe.
Clinical Global Impression (CGI) | Change from Baseline Clinical Global Impression at 6 months.
  The severity of positive, negative, depressive and cognitive symptoms and the overall severity of the disorder will be evaluated. The scale is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients. A higher score indicates a higher severity level.
NEO Five-Factor Inventory | Change from Baseline NEO Five-Factor Inventory at 6 months.
  Measurement of five personality traits: five factors are named Neuroticism (N), Extraversion (E), Openness. Higher scores indicates higher presence of the trait.
  (O), Agreeableness (A), and Conscientiousness (C).
Toronto Alexithymia Scale (TAS) | Change from Baseline Toronto Alexithymia Scale at 6 months.
  Measurement of alexithymia personality trait. Scoring range: 20-100 (higher scores indicate greater impairment).
Global Assessment Functioning (GAF) | Change from Baseline Global Assessment Functioning at 6 months.
  The overall functioning of the patient will be evaluated. The score is between 0-100, where lower scores indicate psychosocial problems that make life difficult for the person under evaluation.
Personal and Social Performance scale (PSP) | Change from Baseline Personal and Social Performance scale at 6 months.
  The specific functioning in 4 main areas will be evaluated. The final score ranges from 100 to 0, where from 100 to 70 points, the ratings refer only to mild difficulties, from 70 to 31 to manifest disabilities of various degrees, and under 30 points, the person's functioning is so poor that intensive support or supervision is needed
EuroQuol-VAS (EQ-VAS) | Change from Baseline EQ-VAS at 6 months.
  Measurement of quality of life according to the patient's perception. It is a 0-100 scale where respondents indicate their overall health status. A higher score indicates higher perceived health.
Boston University Empowerment Scale (BUES) | Change from Baseline Boston University Empowerment Scale at 6 months.
  Measurement of the personal construct of empowerment. The BUES is a 28-item self-report questionnaire which consists of five factors: self-efficacy and self-esteem, power and powerlessness, community activism, righteous anger, and optimism toward and control over the future. Possible scores range from 1 to 4, with higher scores indicating more empowerment.
Questionnaire about the Process of Recovery | Change from Baseline Questionnaire about the Process of Recovery at 6 months.
  Measurement of patient's viewpoint about recovery from psychosis. The QPR is a 15-item self-report questionnaire scored on a 4-point scale (0= disagree strongly, 4=agree strongly). Higher scores are indicative of recovery.
Visual numerical scale of recovery | Change from Baseline Visual numerical scale of recovery at 6 months.
  Subjective measurement of recovery. This scale ranges from 0 to 10, and higher scores are indicative of recovery.
Psychotic Symptom Rating Scales-hallucinations (PSYRATS-H) | Change from Baseline Psychotic Symptom Rating Scales at 6 months.
  Measurement of severity of each hallucination's dimensions. PSYRATS-H is comprised of 11 items on specific dimensions of hallucinations, with each item being rated from 0 (absent) to 4 (severe). The total score ranges from 2 to 44, with higher scores indicating more severe symptoms.
Peters Delusions Inventory (PDI) | Change from Baseline Peters Delusions Inventory at 6 months.
  Assessment of delusional symptoms. The PDI is a 21-item questionnaire. Total score is the sum of positive responses on each item, giving a maximum score of 21 points. Likewise, for each one of the items, there are three subscales that measure degree of conviction, preoccupa- tion, and distress The higher the score, the greater the delusional symptoms is.
Scale Unawareness of Mental Disorders (SUMD) | Change from Baseline Scale Unawareness of Mental Disorders at 6 months.
  Assessment of insight into illness. The scale consists of 3 general items: awareness of mental disorder, awareness of the effects of medication and awareness of the social consequences of the disorder; and of 17 items related to specific symptoms, which make up two subscales: awareness and attribution. Higher scores indicate a lower level of disorder awareness or more incorrect attribution (worse awareness).
Beck Cognitive Insight Scale | Change from Baseline Beck Cognitive Insight Scale at 6 months.
  Assessment of insight into cognitive processes involved in anomalous experiences and misinterpretations. The BCIS is a 15-item self-report questionnaire scored on a 4-point scale (0= do not agree at all, 3= agree completely). It is comprised of two subscales, self-reflectiveness and self-certainty, and a composite Reflectiveness-Certainty Index score. The higher this index score, the greater the cognitive insight is.
Overall Depression Severity and Impairment Scale (ODSIS) | Data will be collected at baseline, throughout the Unified Protocol sessions and immediately after the intervention.
  The level of depression severity will be assessed. ODSIS is a 5-item self-report questionnaire and is scored on a Likert-type scale ranging from 0 to 4. Higher scores indicate greater severity and functional interference associated with depression.
Overall Anxiety Severity and Impairment Scale (OASIS) | Data will be collected at baseline, throughout the Unified Protocol sessions and immediately after the intervention.
  The level of anxiety severity will be assessed. OASIS is a 5-item self-report questionnaire and is scored on a Likert-type scale ranging from 0 to 4. Higher scores indicate greater anxiety-related severity and impairment.
Baron Cohen's Face Test | Data will be collected at the baseline and immediately after the intervention.
  Measurement of capacity to recognise basic and complex emotions in faces. consists of 20-items showing pictures of an actress displaying an emotion. Higher scores indicate a greater capacity for recognizing emotions.
Emotion Regulation Questionnaire (ERQ) | Data will be collected at the baseline and immediately after the intervention.
  Measurement of the tendency to regulate emotions. The ERQ is a self-report questionnaire and is scored on a Likert-type scale, ranging from 1 (strongly disagree) to 7 (strongly agree). It is comprised of two subscales, cognitive reappraisal and expressive suppression. Higher scores indicate higher usage of the strategies.
Difficulties in Emotion Regulation Scale (DERS) | Data will be collected at the baseline and immediately after the intervention.
  Measurement of emotional regulation's dimensions. The DERS is a 28-item self-report questionnaire and is scored on a Likert-type scale, ranging from 1 (almost never) to 5 (almost always). It is comprised of five subscales (inattention, confusion, rejection, interference, lack of control) and a total score. Higher scores indicate higher difficulties in emotion regulation.
Five Facet Mindfulness Questionnaire (FFMQ) | Data will be collected at the baseline and immediately after the intervention.
  Assessment of mindfulness' facets. The FFMQ is a 39-item self-report measure and is scored on a Likert-type scale, ranging from 1 (never) to 5 (very often). It is comprised of five subscales: Observing, Describing, Acting with Awareness, Nonjudging of Inner Experience, and Nonreactivity to Inner Experience. Higher scores represent higher subscale levels of mindfulness.
Involuntary Autobiographical Memory Inventory (IAMI) | Data will be collected at the baseline and immediately after the intervention.
  Measurement of the frequency of involuntary autobiographical memories and involuntary future thoughts. The IAMI is a 20-item self-report measure and is scored on a Likert-type scale, ranging from 0 (never) to 4 (once every hour or more). It is comprised of two subscales: frequency of future involuntary events and frequency of past involuntary events. Higher scores represent higher subscale levels of involuntary memory and thoughts.
Voluntary Control Questions (VCQ) | Data will be collected at the baseline and immediately after the intervention.
  Measurement of the frequency of voluntary autobiographical memories and future thoughts. The VCQ is a 10-item self-report measure and is scored on a Likert-type scale, ranging from 0 (never) to 4 (once every hour or more). It is comprised of two subscales: frequency of future voluntary events and frequency of past voluntary events. Higher scores represent higher subscale levels of voluntary memory and thoughts.
Cognitive Biases Questionnaire for Psychosis (CBQp) | Data will be collected at the baseline and immediately after the intervention.
  Assessment of bias related to psychosis. The CBQp consist of 30 descriptions of everyday situations related to anomalous perceptions or threatening events. Each group of statements covers five cognitive biases: intentionalising, catastrophising, dichotomous thinking, jumping to conclusions and emotional reasoning. Higher scores represent higher level of cognitive biases.
Brief Core Schema Scales | Data will be collected at the baseline and immediately after the intervention.
  Measurement of schemas. The BCSS have 24 items concerning beliefs about the self and others that are assessed on a five-point rating scale (0-4). Four scores are obtained: negative-self, positive- self, negative-others and positive-others. Higher scores indicate a greater endorsement of a schema.
Brief Experiential Avoidance Questionnaire Questionnaire | Data will be collected at the baseline and immediately after the intervention.
  Measurement of the functional process to connect with emotions. The BEAQ is comprised of 15 items, with each item being rated from 1 (Strongly disagree) to 6 (Strongly agree). The total score ranges from 15 to 90, with higher scores indicating more experiential avoidance.

CONTACTS AND LOCATIONS:
Overall Officials: Iluminada Corripio, PhD, Principal Investigator — Hospital de Sant Pau
Locations (1):
- Hospital Santa Creu i Sant Pau, Barcelona, Spain

REFERENCES:
- [Derived] Grasa E, Forment A, Alonso-Solis A, Ramalho L, Roldan A, Pousa E, Ausso S, Berdun J, Genova Tesoro A, Escudero J, Corripio I. Defining the Patient Journey and Identifying Digital Health Solutions in Treatment-Resistant Schizophrenia. Actas Esp Psiquiatr. 2025 Dec;53(6):1208-1222. doi: 10.62641/aep.v53i6.1959. PMID 41437755